CLINICAL TRIAL: NCT04747782
Title: COVID-19 Longitudinal Biomarkers in Lung Injury
Acronym: COLOBILI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Andrew Baker (Other)
Responsible Party: Sponsor-Investigator, Dr. Andrew Baker, Chief, Departments of Critical Care and Anesthesia, St Michael's Hospital, Unity Health Toronto
Organization: Unity Health Toronto (Other)
Other Study IDs: COLOBILI v4.2
Record Dates: First submitted 2021-02-03; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Covid19; Respiratory Disease; Critical Illness
MeSH Terms: conditions — COVID-19; Respiration Disorders; Critical Illness | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * EDTA plasma and cellular pellets, serum, citrated plasma, saliva, fixed whole blood for CYTOF.
  * Percutaneous core biopsy of lung, heart, kidney and muscle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- COVID positive: Patients admitted to the ICU with respiratory distress found to be COVID19 positive.
  Interventions: Other: no interventions performed. Just collecting data, blood samples and post-mortem biopsies.
- COVID negative: Patients admitted to the ICU with respiratory distress found to be COVID19 negative
  Interventions: Other: no interventions performed. Just collecting data, blood samples and post-mortem biopsies.
- COVID positive delayed: Patients admitted to the ICU for an indication other than respiratory distress, found to be COVID19 positive.
  Interventions: Other: no interventions performed. Just collecting data, blood samples and post-mortem biopsies.
- never-ICU: Patients admitted to the internal medicine ward with respiratory distress found to be COVID19 positive.
  Interventions: Other: no interventions performed. Just collecting data, blood samples and post-mortem biopsies.

INTERVENTIONS:
Other: no interventions performed. Just collecting data, blood samples and post-mortem biopsies. — no interventions performed. Just collecting data, blood samples and post-mortem biopsies.

SUMMARY:
Profile known and novel biomarkers in blood in COVID19 patients to characterize the host response to SARS-CoV-2 over time and in response to treatment.

The investigators aim to:

* Better understand the disease. The investigators will achieve this by characterizing the biology of COVID-19 infection and the pathophysiology of the host response using clinical data together with cellular and molecular measurements over the course of the disease. This will allow better insights for the discovery and development of novel therapeutics.
* Understand why different patients have different phenotypes and disease presentations over time. The investigators will achieve this by analyzing for patient subgroups. This will allow targeted patient stratification and better matching of resources.
* Understand how patients are responding to the different medications being tested in clinical trials. The investigators will achieve that by co-enrolling with therapeutic trials. This will allow an understanding of the biological effects of these interventions.

Study Design: Observational adaptive study of a translational nature, combining clinical data and basic science investigations in blood samples in the same patients, longitudinally, with serial interim analyses.

Primary outcomes: 90 day ICU mortality. Secondary outcomes: measures of ICU utilization and disease severity, and 90 day in-hospital mortality.

The study ends after 3 months from admission to the ICU, hospital discharge or death.

Location: St. Michael's Hospital (Unity Health Toronto), an academic center in downtown Toronto affiliated with the University of Toronto.

The investigators will collect: A) Detailed clinical data including investigations, mechanical ventilation and cardiovascular parameters. B) Blood samples for state-of-the-art multi-omics biomarker discovery and development: cytokines, anti-COVID19 antibodies, autoimmune serology, metabolomics, transcriptomics, epigenomics, deep immune phenotyping, viral loads. For those patients who die with COVID19 The investigators will perform bedside post-mortem biopsies of lung, heart, kidney and muscle.

Sampling times: From admission to the maximal severity phase through convalescence, in order to capture the evolution and dynamics of the disease and the recovery process: days 0,1, 3, 5, 7, 10, 15 and 22, and then every 2 weeks until the end of the study (3 months from admission to the ICU, hospital discharge or death).

ELIGIBILITY:
* Primary Cohort: Patients admitted to the ICU with respiratory deterioration suspected or confirmed to be due to SARS-CoV-2. Suspicion will be based on the clinical criteria in place at SMH, with the threshold for inclusion being a suspicion high enough to use PPE until confirmatory testing results are obtained. Only patients found to be COVID19 positive will stay in this cohort. This population will be called "ICU Positive".
* Secondary Cohort: Patients admitted to the ICU for any reason who are COVID19 positive, regardless of admission date or when they are found to be COVID19 positive. This population will be called "ICU Positive - delayed"
* Biological controls in the ICU: Any patients from the primary cohort who are found to be COVID19 negative. This population will be called "ICU negative".
* Biological controls outside the ICU: Patients admitted to the floor with respiratory deterioration suspected or confirmed to be due to SARS-CoV-2, or that develop such respiratory deterioration within 15 days of admission (i.e. become "persons under investigation"). Suspicion will be based on the clinical criteria in place at SMH, with the threshold for inclusion being a suspicion high enough to use PPE until confirmatory testing results are obtained. Only patients found to be COVID19 positive will stay in this cohort. If these patients require ICU admission within 15 days, they will cross-over to the "ICU positive" cohort and count towards that cohort (i.e. number of recruited patients). If they don't require ICU admission within 15 days, they will stay in this cohort and be called "never ICU".
* Healthy volunteers: The investigators will recruit healthy volunteers among healthcare workers and allied personnel in the hospital. They will provide peripheral blood to serve as: a) independent controls for experimental and laboratory variables, and b) references of healthy baseline state for experiments.
* A patient previously enrolled as a COVID negative can be re-enrolled in a subsequent hospitalization with a new study ID (i.e. counts as another encounter for the total enrollment). The records will be linked to indicate they represent the same person enrolled again.

Exclusion Criteria

* Refusal to participate.
* Inability to record the primary outcome during the first 2 weeks.
* For the ICU positive and ICU negative cohorts only: failure to obtain the day 0 or 1 blood sample (for example technical problems, or identification of COVID-19 after ICU admission i.e. there was no suspicion on admission).
* For the ward patients, inability to collect day 1 or 2 blood sample.
* Known to have had COVID in the past (>4 weeks) in any setting.
* Healthy volunteers only: COVID19 known or suspected infection, or unprotected exposure to a known acutely ill COVID19 patient in the past 4 weeks; and/or currently unwell or in the course of an acute illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the critical care unit or general medicine ward in a tertiary referral medical center.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-03-23 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Death in ICU | within 3 months from admission
  Death in ICU

SECONDARY OUTCOMES:
Days in ICU | within 3 months from admission to the ICU
  Length of hospitalization
Mechanical ventilation days | within 3 months from admission to the ICU
  Length of mechanical ventilation while in the ICU
Days of mechanical ventilation rescue measures | within 3 months from admission to the ICU
  Number of days on which the patient was treated with one or more of the following rescue meaures: neuromuscular blockade, inhaled NO, proning.
APACHE II score on admission | On admission to the ICU
  Acute Physiology And Chronic Health Evaluation II. Min 0, Max 71. Higher scores impart higher mortality risk.
SOFA score | On the same days as blood sampling: days 0,1, 3, 5, 7, 10, 15 and 22, and then every 2 weeks until the end of the study (3 months from admission to the ICU, hospital discharge or death).
  Sequential Organ Failure Assessment, calculated daily. Min 6, Max 24. Higher scores impart higher mortality risk.
In hospital death | within 3 months from admission
  In hospital death

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Baker, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Depends on the type of data requested

REFERENCES:
- [Derived] Trahtemberg U, Fritzler MJ; On behalf of the COVID-19 chapter of the "Longitudinal Biomarkers in Lung Injury" study group. COVID-19-associated autoimmunity as a feature of acute respiratory failure. Intensive Care Med. 2021 Jul;47(7):801-804. doi: 10.1007/s00134-021-06408-z. Epub 2021 Apr 30. No abstract available. PMID 33928414
- [Derived] Trahtemberg U, Rottapel R, Dos Santos CC, Slutsky AS, Baker A, Fritzler MJ. Anticardiolipin and other antiphospholipid antibodies in critically ill COVID-19 positive and negative patients. Ann Rheum Dis. 2021 Sep;80(9):1236-1240. doi: 10.1136/annrheumdis-2021-220206. Epub 2021 Apr 26. PMID 33903092